CLINICAL TRIAL: NCT00558987
Title: Enhancing Anticipatory Guidance About Discipline for Low-Income Families: A Video Intervention Project
Brief Title: Parenting Videos In Primary Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: The Thomas Wilson Sanitarium for Children of Baltimore City (Other)
Responsible Party: Anne Duggan, ScD, Johns Hopkins University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: TW-101251; NA_00012021
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Discipline Attitudes; Discipline Practices
Keywords: Discipline; Parenting; Primary Care; Videos

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental)
  Interventions: Behavioral: Discipline Video
- 2 (Sham Comparator)
  Interventions: Behavioral: Nutrition Video

INTERVENTIONS:
Behavioral: Discipline Video — 1. The discipline video will be shown to the caregiver before the visit while they are waiting to see the doctor. The video gives specific guidance on avoiding physical discipline, setting consistent, safe and age appropriate limits.
  2. A copy of the discipline video and the handout reinforcing the messages presented in the video will be given to the caregiver by the research staff to share with other caregivers.
  Other Names: "Positive discipline: Vol. 2" by Injoy Videos
  Arms: 1
Behavioral: Nutrition Video — A brief educational video on nutrition information, a topic not related to discipline.
  Other Names: "Childhood Nutrition: Vol. 2" by Injoy Videos
  Arms: 2

SUMMARY:
The purpose of this study is to test the effectiveness of a video-based parent education intervention delivered in the primary care setting on parents and other caregivers discipline attitudes and practices.

ELIGIBILITY:
Inclusion Criteria:

* Adult caregivers of children ages 12 to 36 months with a scheduled well-child visit.
* Caregivers must be older than 18 years of age, must be considered a consistent caregiver for the child, must be the primary caregiver at least 2 days per week, and must live with the child.

Exclusion Criteria:

* Caregivers previously enrolled in the study.
* Caregivers who do not speak or read English,
* Caregivers not able to give contact information for follow-up,
* Caregivers of a child who has a severe behavioral problem or developmental delay as reported by the parent during the initial recruitment phone call.

Min Age: 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2008-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Frequency of spanking | baseline and 6 week follow-up

SECONDARY OUTCOMES:
Attitudes about Discipline | baseline and 6 week follow-up
Type of discipline practices used | baseline and 6 week follow-up
Discussion with pediatric provider | immediately post visit

CONTACTS AND LOCATIONS:
Overall Officials: Rachel A Dodge, MD, MPH, Study Director — Johns Hopkins University; Anne K Duggan, ScD, Principal Investigator — Johns Hopkins University
Locations (1):
- Harriet Lane Primary Care Clinic, Baltimore, Maryland, United States